CLINICAL TRIAL: NCT02840435
Title: Pilot Study on Mindfulness Training for Smokers Via Web-based Video and Telephone Counseling
Brief Title: Study on Sit to Quit Phone Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Consumer Wellness Solutions (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00073392; P50DA027840 (NIH)
Record Dates: First submitted 2016-07-05; First posted 2016-07-21 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Nicotine Dependence
Keywords: Nicotine addiction; Cigarette smoking
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- North Carolina Quit Line: Quit for Life (Active Comparator): Participants will be connected to the 'Quit for Life' program offered through the North Carolina Quit Line.
  Interventions: Behavioral: Quit for Life
- Sit to Quit (Experimental): Participants will be connected to the 'Sit to Quit' program offered through the Duke Smoking Cessation Program.
  Interventions: Behavioral: Sit to Quit

INTERVENTIONS:
Behavioral: Sit to Quit — Sit to Quit(STQ) is a smoking cessation program adapted from Mindfulness Training for Smokers (MTS) with core content available on the STQ video. STQ contains many elements found in traditional interventions (e.g. instruction on planning and structuring a quit day, garnering support from others, assessment of prior relapse occasions, development of strategies to avoid triggers). In addition, STQ provides instruction in various mindfulness practices and in how to apply mindfulness skills to manage common causes of relapse. Exercises are provided, and it is recommended to learn the skill experientially. STQ requests that participants practice guided meditation each day using an audio recording and employ other mindfulness practices targeted to manage relapse challenges. Participants will also receive the STQ Participant Manual, which provides all the instruction found in the STQ Video, but provides additional discussion of topics for smokers who desire additional material.
  Other Names: Mindfulness Training for Smokers
  Arms: Sit to Quit
Behavioral: Quit for Life — Quit for Life integrates telephone counseling, written materials, NRT, and an online program called "Web Coach." Web Coach is an interactive internet-based support system that provides health information on smoking cessation, assistance in the development of quit strategies, and an interactive blog to interact with other smokers. Web Coach is used by approximately 70% of AWI callers. Web Coach is not a complete program, but instead is designed to supplement AWI phone-based therapy. In addition, Quit for Life also provides the "Quit Guide," which is a smoking cessation manual with written instructions on the use of medications, planning a quit day, and cessation-related cognitive skills.
  Other Names: North Carolina Quit Line
  Arms: North Carolina Quit Line: Quit for Life

SUMMARY:
This study is designed to test the effectiveness of the smoking cessation intervention "Sit to Quit" through a randomized-control trial. This study will compare abstinence outcomes in the Sit to Quit study group to a control group using the North Carolina State Tobacco Quit Line.

DETAILED DESCRIPTION:
This study is designed to test the effectiveness of the smoking cessation intervention "Sit to Quit" through a randomized-control trial. This study will compare abstinence outcomes in the Sit to Quit study group to a control group using the North Carolina State Tobacco Quit Line. This is an investigational study (n=60) designed to test Sit to Quit (STQ) versus Quit Line (QL) through a pilot randomized control trial. The proposed study is designed with double-blind procedures (participants and study staff) for randomization of 60 participants recruited through Duke Smoking Cessation Program into two groups: STQ and QL. STQ participants will receive access to the STQ Instructional Video, the STQ manual, and proactive Quit Coach calls supporting STQ. QL participants will be instructed to contact the NC Quit Line and will receive access to "web Coach" (Alere Well-being site), the Quit Line manual, and proactive Quit Coach calls supporting "Quit for Life." All statistical analysis will be performed under the directions of the statistician designated in key personnel. Outcomes of variables including: demographic variables, evaluation responses, and abstinence rates will be analyzed using general regression models using an ANOVA-based design. The study Principal Investigator Dr. James Davis will ultimately be responsible for data and safety monitoring. Subject data will be collected during visits and captured in the Electronic Medical Record. Data will be collected by phone, and this data will be stored in REDCap. Participants that experience events related to their clinical treatment will be recommended to follow-up with their provider.

ELIGIBILITY:
Inclusion Criteria:

* Patient being treated at Duke Smoking Cessation Program for tobacco use
* Age 18 years or older
* Actively smoking 5 or more cigarettes per day for at least one year
* Fluency in spoken and written English
* Willing to set a quit date within 2 weeks
* Access to a smart phone or internet and telephone
* Willingness to watch 3 videos on computer, receive 5 counseling calls, and attend investigational visits.

Exclusion Criteria:

* CO test under 7 ppm during initial screening
* 8 or above on the Alcohol Use Disorders Identification Test (AUDIT-10)
* 6 or above on Drug Abuse Screening Test (DAST-10)
* 3 or above on Patient Health Questionnaire (PHQ-2) Depression Scale
* Daily use of a second form of tobacco or nicotine (e.g. e-cigarettes, cigars, chewing tobacco, snuff)
* Current use of a smoking cessation medication (e.g. nicotine replacement, Varenicline, Bupropion)
* Intolerable side effects related to, refusal to take, or medical contraindication with nicotine patch
* Symptomatic cognitive or emotive disorder such as untreated schizophrenia, severe untreated depression, or severe untreated anxiety. This is determined by clinical assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Biochemically confirmed continuous 30-day abstinence from smoking | 12 weeks post-Target Quit Day (TQD)
  Biochemically confirmed 30-day continuous abstinence. Abstinence is determined by a participant both reporting not smoking in the past 30 days AND a result of < 7 ppm in carbon monoxide breath testing. If the participant does not meet both criteria, they are not considered abstinent

SECONDARY OUTCOMES:
Biochemically confirmed 7-day point prevalence abstinence from smoking | 12 weeks post-TQD
  Biochemically confirmed 7-day continuous abstinence. Abstinence is determined by a participant both reporting not smoking in the past 7 days AND a result of < 7 ppm in carbon monoxide breath testing. If the participant does not meet both criteria, they are not considered abstinent
Biochemically confirmed 7-day point prevalence abstinence from smoking | 2 weeks post-TQD
  Biochemically confirmed 7-day continuous abstinence. Abstinence is determined by a participant both reporting not smoking in the past 7 days AND a result of < 7 ppm in carbon monoxide breath testing. If the participant does not meet both criteria, they are not considered abstinent
Self-reported 7-day point prevalence abstinence rates | 1 week post TQD
  7-day point prevalence abstinence as measured by phone-based, single-item self-report
Self-reported 7-day point prevalence abstinence rates | 12 weeks post TQD
  7-day point prevalence abstinence as measured by phone-based, single-item self-report
Self-reported 7-day point prevalence abstinence rates | 26 weeks post TQD
  7-day point prevalence abstinence as measured by phone-based, single-item self-report
Self-reported 7-day point prevalence abstinence rates | 6 weeks post TQD
  7-day point prevalence abstinence as measured by phone-based, single-item self-report
Self-reported 7-day point prevalence abstinence rates | 2 weeks post TQD
  7-day point prevalence abstinence as measured by phone-based, single-item self-report
Smoking reduction | 1 week post-TQD
  Smoking reduction as measured by number of cpd measured by phone-based self-report
Smoking reduction | 2 weeks post-TQD
  Smoking reduction as measured by number of cpd measured by phone-based self-report
Smoking reduction | 6 weeks post-TQD
  Smoking reduction as measured by number of cpd measured by phone-based self-report
Smoking reduction | 12 weeks post-TQD
  Smoking reduction as measured by number of cpd measured by phone-based self-report
Smoking reduction | 26 weeks post-TQD
  Smoking reduction as measured by number of cpd measured by phone-based self-report
Changes in stress | Baseline to 2-week and 12-week post TQD
  Change in self-reported measures of stress
Changes in anxiety | Baseline to 2-week and 12-week post TQD
  Change in self-reported measures of anxiety
Changes in depression | Baseline to 2-week and 12-week post TQD
  Change in self-reported measures of depression
Changes in relapse predictors | Baseline to 1-week post-TQD, 2-week post-TQD, 6-week post-TQD, 12-week post-TQD, and 26-week post-TQD
  Changes in self-reported measures on repeated non-standardized single-item question on stress, urges, and confidence assessed by phone
Feasibility: attendance records | Up to 12 weeks post-TQD
  Feasibility as measured by attendance and completion of STQ and QL assessed by attendance records taken instructors during phone sessions.
Feasibility: website usage | Up to 12 weeks post-TQD
  Feasibility as measured by website usage by electronically recording login and using a site-based timer to record time accessing the site through each intervention
Feasibility: course evaluation | Up to 12 weeks post-TQD
  Feasibility as measured by course evaluation
Feasibility: demographics | 12-weeks post-TQD
  Feasibility as measured by demographics of patients at DSCP
Feasibility: Behavioral intervention used | 12 weeks post-TQD
  Feasibility as measured by behavioral intervention assignment
Feasibility: Attendance at DSCP appointments | 12 weeks post-TQD
  Feasibility as measured by attendance at DSCP appointments
Feasibility: Referral routes to DSCP | Baseline
  Feasibility as measured by referral routes to DSCP
Feasibility: Side effects | 1-week post-TQD, 2-week post-TQD, and 6-week post-TQD
  Feasibility as measured by side effects, as measured by phone assessment
Feasibility: medication adherence | 1-week post-TQD, 2-week post-TQD, 6-week post-TQD, and 26-week post-TQD
  Feasibility as measured by medication adherence, as measured by phone assessment
Feasibility: mindfulness practices | 1-week post-TQD, 2-week post-TQD, 6-week post-TQD, and 26-week post-TQD
  Feasibility as measured by non-standardized phone-based self-report of number of times mindfulness practices are used by experimental group
Feasibility: meditation time | 1-week post-TQD, 2-week post-TQD, 6-week post-TQD, and 26-week post-TQD
  Feasibility as measured by non-standardized phone-based self-report of time spent meditating by experimental group

CONTACTS AND LOCATIONS:
Overall Officials: James M Davis, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center for Smoking Cessation, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No